CLINICAL TRIAL: NCT03044587
Title: Nal-IRI With 5-fluorouracil (5-FU) and Leucovorin or Gemcitabine Plus Cisplatin in Advanced Biliary-tract Cancer - An Open Label, Non-comparative, Randomized, Multicenter Phase II Trial
Brief Title: Nal-IRI With 5-fluorouracil (5-FU) and Leucovorin or Gemcitabine Plus Cisplatin in Advanced Biliary-tract Cancer
Acronym: NIFE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Servier (Industry); Institut für Klinisch-Onkologische Forschung der Krankenhaus Nordwest GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-YMO/HEP-0315; 2016-002467-34 (EudraCT Number); O16-33004 (Other: Baxalta GmbH)
Record Dates: First submitted 2017-01-23; First posted 2017-02-07 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Adenocarcinoma Metastatic; Biliary Tract Cancer; Adenocarcinoma of the Biliary Tract; Adenocarinoma Locally Advanced; Non-Resectable Hepatocellular Carcinoma; Intrahepatic Bile Duct Carcinoma; Extrahepatic Bile Duct Carcinoma
Keywords: Biliary Tract Cancer; NaI-IRI
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Bile Duct Neoplasms | interventions — Fluorouracil; Leucovorin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm NaI-IRI + 5-FU + Leucovorin (Arm A) (Experimental): Nal-IRI [Irinotecan liposome], 5-FU [5-Fluorouracil], Leucovorin Cycle q2w
  Interventions: Drug: Arm NaI-IRI + 5-FU + Leucovorin (Arm A)
- Arm Cisplatin + Gemcitabine (Arm B, standard of care) (Other): Cisplatin, Gemcitabine Cycle q3w
  Interventions: Drug: Arm Cisplatin + Gemcitabine (Arm B)

INTERVENTIONS:
Drug: Arm NaI-IRI + 5-FU + Leucovorin (Arm A) — Nal-IRI (80 mg/m2 as a 1.5 hour infusion), 5-FU (2400 mg/m2 as 46 hour infusion) and Leucovorin (400 mg/m2 as 0.5 hour infusion) Cycle q2w
  Arms: Arm NaI-IRI + 5-FU + Leucovorin (Arm A)
Drug: Arm Cisplatin + Gemcitabine (Arm B) — Cisplatin (25 mg/m2 as 1 hour infusion on D1, D8) and Gemcitabine (1000 mg/m2 as 0.5 hour infusion on D1, D8) Cycle q3w
  Arms: Arm Cisplatin + Gemcitabine (Arm B, standard of care)

SUMMARY:
AIO-YMO/HEP-0315 (NIFE) is an open label, non-comparative, randomized, multicenter phase II trial

DETAILED DESCRIPTION:
The primary objective is to determine whether a combination of 5-FU and nal-IRI prolongs progression-free survival in patients with locally advanced or metastatic adenocarcinoma of the biliary tract

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent incl. participation in translational research and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age ≥ 18 years at time of study entry
3. Histologically confirmed, non-resectable, locally advanced or metastatic adenocarcinoma of the intrahepatic or extrahepatic biliary tract
4. Protocol-specific staging guidelines have to be observed and non-resectability has to be confirmed by local tumor board
5. Measurable or assessable disease according to RECIST 1.1
6. ECOG performance status 0-1
7. Life expectancy of more than 3 months
8. If applicable, adequately treated biliary tract obstruction before study entry with total bilirubin concentration ≤ 2 x ULN
9. Adequate blood count, liver-enzymes, and renal function:

   * White blood cell count ≥ 3.5 x 10^6/mL
   * Platelet count ≥ 100 x 10^9/L (>100,000 per mm3)
   * AST (SGOT)/ALT (SGPT) ≤ 5 x institutional upper limit of normal
   * Serum Creatinine ≤ 1.5 x ULN and a calculated glomerular filtration rate ≥ 30 mL per minute
10. Patients not receiving therapeutic anticoagulation must have an INR < 1.5 ULN and PTT < 1.5 ULN within 7 days prior to randomization. The use of full dose anticoagulants is allowed as long as the INR or PTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least three weeks at the time of randomization
11. No prior palliative chemotherapy for biliary tract cancer
12. No adjuvant treatment within 6 months prior to study entry
13. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Active uncontrolled infection, chronic infectious diseases, immune deficiency syndromes
2. Premalignant hematologic disorders, e.g. myelodysplastic syndrome
3. Clinically significant cardiovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) within 6 months before enrollment
4. Prior (>5 years) or concurrent malignancy (other than biliary-tract cancer) which either progresses or requires active treatment. Exceptions are: basal cell cancer of the skin, pre-invasive cancer of the cervix, T1a or T1b prostate carcinoma, or superficial bladder tumor [Ta, Tis and T1].
5. Pre-existing lung disease
6. History or clinical evidence of CNS metastases

   Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria:
   1. are asymptomatic and
   2. have no requirement for steroids 6 weeks prior to start of study treatment. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS metastases
7. History of hypersensitivity to any of the study drugs or any of the constituents of the products
8. Allogeneic transplantation requiring immunosuppressive therapy or other major immunosuppressive therapy
9. Severe non-healing wounds, ulcers or bone fractions
10. Evidence of bleeding diathesis or coagulopathy
11. Major surgical procedures, except open biopsy, nor significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgical procedure during the course of the study except for surgery of central intravenous line placement for chemotherapy administration.
12. Medication that is known to interfere with any of the agents applied in the trial.
13. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessary (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (serum β-HCG) at Screening.
14. Known Gilbert-Meulengracht syndrome
15. Known chronic hypoacusis, tinnitus or vertigo
16. Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
17. Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is of longer duration.
18. Previous enrollment or randomization in the present study (does not include screening failure).
19. Any other chemotherapy at study start
20. Involvement in the planning and/or conduct of the study
21. Patient who might be dependent on the sponsor, site or the investigator
22. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities.
23. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival [PFS] | approx. 25 months

SECONDARY OUTCOMES:
Overall progression free survival according to RECIST 1.1 | approx. 54 months
  Response Evaluation Criteria in Solid Tumors (RECIST 1.1.)
3-years overall survival | approx. 36 months
  3-years overall survival
Disease control rate according to RECIST 1.1 | approx. 54 months
Objective tumor response rate (ORR) according to RECIST 1.1 | approx. 54 months
  Proportion of patients with an objective response according to RECIST 1.1
Toxicity/Safety according to CTC-AE-criteria | approx. 54 months
Health related quality of life | approx. 54 months
  EORTC QLQ-BIL21
Health related quality of life | approx. 54 months
  EORTC QLQ-C30
Health related quality of life | approx. 54 months
  Hospital Anxiety and Depression Scale (HADS-D)
Retrospective correlation of resectability in accordance with a central surgical board compared to local surgical review | approx. 54 months
  Tumor resectability in accordance with a retrospective central surgical board compared to local surgical review
Retrospective central radiological review | approx. 54 months

OTHER OUTCOMES:
Exploratory biomarkers analysis | approx. 54 months
  cfDNA exome sequencing, transcriptome, miRNA-arrays prior to and after start of treatment and upon progress
Establishment of Predictive/Prognostic biomarker profiles for advanced cholangiocarcinoma | approx. 54 months
Tumor Evolution under systemic therapy | approx. 54 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Ettrich, Dr., Principal Investigator — Klinik für Innere Medizin I, Universitätsklinikum Ulm
Locations (1):
- Universitätsklinikum Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ettrich TJ, Modest DP, Sinn M, Striefler JK, Opitz B, Goetze T, Gallmeier E, Angermeier S, Fischer von Weikersthal L, Jacobasch L, Waldschmidt D, Niedermeier M, Sohm M, Berger AW, Manzini G, Fehrenbach U, Auer TA, Hosse C, Vogele D, Sookthai D, Schaaf M, Muche R, Hinke A, Seufferlein T, Perkhofer L. Nanoliposomal Irinotecan With Fluorouracil and Leucovorin or Gemcitabine Plus Cisplatin in Advanced Cholangiocarcinoma: A Phase II Study of the AIO Hepatobiliary-YMO Cancer Groups (NIFE-AIO-YMO HEP-0315). J Clin Oncol. 2024 Sep 10;42(26):3094-3104. doi: 10.1200/JCO.23.01566. Epub 2024 Jun 6. PMID 38843469
- [Derived] Perkhofer L, Berger AW, Beutel AK, Gallmeier E, Angermeier S, Fischer von Weikersthal L, Goetze TO, Muche R, Seufferlein T, Ettrich TJ. Nal-IRI with 5-fluorouracil (5-FU) and leucovorin or gemcitabine plus cisplatin in advanced biliary tract cancer - the NIFE trial (AIO-YMO HEP-0315) an open label, non-comparative, randomized, multicenter phase II study. BMC Cancer. 2019 Oct 23;19(1):990. doi: 10.1186/s12885-019-6142-y. PMID 31646981
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de
- See also: AIO-Studien-gGmbH — http://www.aio-studien-ggmbh.de